CLINICAL TRIAL: NCT01576835
Title: Comparison of Non-contrast Renal Artery Magnetic Resonance Angiography With Contrast-enhanced CT Angiography
Brief Title: Renal Artery Contrast-Free Trial
Acronym: REACT
Status: Completed | Type: Observational
Sponsor: Central Coast Cardiovascular Research (Other)
Collaborators: Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Timothy Albert MD, FACC, Secretary, Central Coast Cardiovascular Research
Other Study IDs: REACT2012
Record Dates: First submitted 2012-04-10; First posted 2012-04-13 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Renal Artery Stenosis; Kidney Diseases; Hypertension
Keywords: Non-contrast
MeSH Terms: conditions — Renal Artery Obstruction; Kidney Diseases; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will compare the results of a clinically ordered abdominal CT angiography to a research non-contrast MR angiogram (MRA). CTA is a "gold-standard" for identifying blockages in the kidney arteries or other blood vessel problems. CTA requires radiation and contrast to obtain useful images. Conversely, the MR abdomen technique being used for the study uses no radiation or contrast and is felt to be a safer option for individuals who have kidney problems. there is benefit to establishing non-contrast MRA as a clinically accurate test.

DETAILED DESCRIPTION:
REACT is a prospective, minimal-risk, and multi-center international trial. The purpose of the study is to evaluate the safety and efficacy of non-contrast magnetic resonance angiography (MRA) for the diagnosis of renal artery stenosis (RAS).

The current "gold standards" for diagnosing RAS are non-invasive 3D angiography with contrast-enhanced CTA/MRA or invasive X-ray angiography. All of these techniques require the use of an intravenous injection of either iodinated contrast material or gadolinium based agents.

Iodinated contrast agents are contraindicated in patients with renal dysfunction and have increased risk of allergic reaction. Contrast-enhanced magnetic resonance angiography (MRA) with gadolinium has fewer risks associated with it, however, is currently contraindicated in patients with severe renal insufficiency because of concerns about developing a rare but often fatal condition termed nephrogenic systemic fibrosis (NSF).

Non-contrast MRA techniques are felt to provide an avenue for safer, effective vascular imaging in patients both with and without kidney dysfunction. In this trial we propose to validate the contrast-free MRA technique, T-SLIP (time-spatial labeling inversion pulse), for diagnosing RAS. This study will compare T-SLIP to the reference standard of contrast-enhanced CTA and is designed to test its efficacy, reproducibility, reliability, and safety.

ELIGIBILITY:
Inclusion Criteria:

* The abdominal CTA evaluation form has been completed and confirmed to fit criteria for study enrollment
* The research MRA will be completed within 3 months of abdominal CTA
* Subject signed and dated the informed consent form
* Subject agrees to a "research" abdominal MRA
* Subject is able to follow breathing and scanning instructions
* Subject is at least 18 years of age

Exclusion Criteria:

* Subject has had a significant change in clinical condition between the time of abdominal CTA and abdominal MRA (e.g. worsening renal function, renal vascular intervention)
* Subject has renal stents, or other known material that may affect MR image quality
* Subject has a contraindication to an MRI
* Subject had intravenous gadolinium media within the previous 24 hours
* Subject has a baseline heart rate >90 beats per minute or respiratory rate >25 breaths/minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have had an abdominal CT for any reason will be considered for the REACT study. They may be referred from private practice or imaging center.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of non-contrast renal MR angiography for assessment of renal artery stenosis (RAS) | up to study closure, estimated 3 months
  Accuracy of renal T-SLIP for assessing RAS severity in comparison to abdominal CTA. CTA is being used as the gold standard for comparison

SECONDARY OUTCOMES:
Safety assessment of non-contrast renal artery imaging | may be followed on average up to 3 months after closure
  Safety assessment of T-SLIP will be reported by documenting adverse clinical events (e.g. patient discomfort during scan)
Image quality | up to study closure, estimated 3 months
  MR angiography image quality will be determined in a blinded fashion by two independent readers. This will be reported separately.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S. Albert, MD, Principal Investigator — Central Coast Cardiovascular Research
Locations (1):
- Central Coast Cardiolgy, Salinas, California, United States